CLINICAL TRIAL: NCT03093922
Title: Atezolizumab in Combination With Gemcitabine and Cisplatin As First-Line Treatment in Metastatic Urothelial Cancer: A Multicenter Randomized Phase II Study of Two Alternative Dosing Schedules
Brief Title: A Study of Two Dosing Schedules of Atezolizumab in Combination With Gemcitabine and Cisplatin as First-Line Treatment for Metastatic Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ohio State University (Other); University of Chicago (Other); Genentech, Inc. (Industry); Targos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1621
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Carcinoma; Locally Advanced; Unresectable
Keywords: Gemcitabine; Atezolizumab; Cisplatin; 16-1621
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a randomized phase II study testing two different schedules of atezolizumab combined with gemcitabine and cisplatin chemotherapy (GC) in patients with metastatic urothelial carcinoma (mUC) who are eligible for cisplatin.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atezolizumab alone with Gemcitabine and Cisplatin (Experimental): Atezolizumab alone for 2 cycles. One treatment cycle equals 21 days. Then patient will receive combined atezolizumab and Gemcitabine and Cisplatin for 6 cycles. All 8 treatment cycles will take approximately 24 weeks. If carboplatin is substituted for cisplatin, eGFR for dosing may be calculated by institutional standard formulas, at the discretion of the treating investigator. This cohort is NO LONGER ACCRUING patients since 5/22/2018.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Cisplatin
- Atezolizumab with Gemcitabine and Cisplatin (Experimental): Gemcitabine and Cisplatin for 2 cycles. One treatment cycle equals 21 days. After 2 cycles of Gemcitabine and Cisplatin patient will receive combined atezolizumab and Gemcitabine and Cisplatin for 4 cycles. All 6 treatment cycles will take approximately 18 weeks. If carboplatin is substituted for cisplatin, eGFR for dosing may be calculated by institutional standard formulas, at the discretion of the treating investigator.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Cisplatin
- Atezolizumab alone for 1 cycle prior to gemcitabine, cisplatin (Experimental): Atezolizumab alone for 1 cycle. One treatment cycle equals 21 days. After 1 cycle of atezolizumab the patients will receive combined atezolizumab and gemcitabine, cisplatin for 4 cycles. All 5 treatment cycles will take approximately 15 weeks. Cisplatin dose can be given on day 1 or split over days 1 and 8 at the investigator"s discretion. Once the split-dose cisplatin is used, it should be used for the remainder of the chemotherapy treatment course.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg/m^2
Drug: Gemcitabine — 1000 mg/m^2
Drug: Cisplatin — 70 mg/m^2

SUMMARY:
The purpose of this study is to compare any good and bad effects the study drug atezolizumab has on the cancer when combined with the standard chemotherapy drugs gemcitabine and cisplatin (or GC) in two different dosing schedules: chemotherapy (GC) before atezolizumab vs. GC after atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed urothelial carcinoma of the bladder, ureter, urethra, or renal pelvis by the enrolling institution. Patients with mixed histologies are required to have a predominant urothelial component as reviewed by the pathologist at the enrolling institution.
* Locally advanced (T4b, any N: any T, N2-3) or metastatic (M1) disease as determined by the treating investigator.
* Age ≥18 years
* Life expectancy ≥ 12 weeks
* The patient must have measurable disease according to RECIST v1.1 and must have one site amenable to biopsy that, in the opinion of the investigator and/or interventional radiologist, is likely to yield acceptable tumor sample for a core biopsy per the below pathology criteria.
* Subject must agree to undergo two research-directed biopsies during treatment.
* Patients must have adequate tumor tissue available for PD-L1 testing. Adequate tumor tissue is defined as:

  * For core-needle biopsy specimens, at least three cores should be submitted for evaluation if feasible. Acceptable samples include core-needle biopsies for deep tumor tissue (minimum of three cores) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions. Samples collected from fine-needle aspiration, brushing, cell pellet from pleural effusion, bone metastases without a soft tissue component, and lavage are not acceptable.
  * For pre-treatment archival tissue, representative urothelial carcinoma FFPE tumor specimens (tumor blocks or 30 unstained slides) must be provided. Patients with < 30 slides may be enrolled after discussion with the MSK Principal Investigator.
  * Primary or metastatic specimens (with the exception of bone because it is not evaluable for PD-L1 expression) may be submitted.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1):

  * ANC ≥ 1500 cells/uL
  * WBC counts > 2500/uL
  * Lymphocyte count ≥ 300/uL
  * Platelet count ≥ 100,000/uL; Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception:
  * Patients with known Gilbert disease who have total bilirubin level ≤ 3 x ULN may be enrolled.
* AST and ALT ≤ 3.0 x ULN with the following exception:

  °Patients with liver metastases may enroll with AST and ALT ≤ 5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN with the following exception:

  °Patients with documented liver or bone metastases may enroll with alkaline phosphatase ≤ 5 x ULN
* Estimated glomerular filtration rate (eGFR) ≥ 50 ml/min/1.73m^2 using the CKD-EPI equation: eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of --Scr/k or 1, and max indicates the maximum of Scr/k or 1
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 5 months after the last dose of atezolizumab.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* INR and aPTT ≤ 1.5 x ULN

  * This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.
* Ability and willingness to comply with the requirements of the study protocol

Exclusion Criteria:

* Prior chemotherapy or immunotherapy for metastatic urothelial cancer. Prior neoadjuvant or adjuvant chemotherapy with first progression > 12 months is allowed. Prior intravesical treatments such as BCG are allowed, however no BCG is allowed within 4 weeks prior to initiation of study treatment.
* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to Cycle 1, Day 1. Herbal therapy intended as anticancer therapy must also be discontinued at least 1 week prior to Cycle 1, Day 1.
  * Palliative radiotherapy for bone metastases > 2 weeks prior to Cycle 1, Day 1
* Bisphosphonate therapy for symptomatic hypercalcemia

  °Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Patients with a history of or active bone marrow disorders expected to interfere with study therapy (e.g. acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma)
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases

  * Evaluable or measurable disease outside the CNS
  * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
  * No history of intracranial hemorrhage or spinal cord hemorrhage
  * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.
  * No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1
* Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1, Day 1 Screening CNS radiographic study ≥ 4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids

* Pregnancy, lactation, or breastfeeding.
* Evidence of NYHA functional class III or IV heart disease
* Sensory or motor peripheral neuropathy ≥ grade 2
* Hearing loss ≥ grade 2
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. The following are exceptions to this criterion.

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Patients with celiac disease controlled on diet alone may be eligible
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (i.e. not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  °History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1 °Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study

  °Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as but not limited to adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.)
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

  °Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met: Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose No history of severe immune-related adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4)
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half-lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 year
  with response determined according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Funt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Ohio State University, Columbus, Ohio

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm